CLINICAL TRIAL: NCT00802373
Title: Solifenacin in a Flexible Dose Regimen With Tolterodine as an Active Comparator in a Double-blind, Double-dummy, Randomised Overactive Bladder Symptom Trial
Brief Title: Solifenacin Succinate Versus Tolterodine 4mg Once Daily
Acronym: STAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 905-EC-001
Record Dates: First submitted 2008-12-02; First posted 2008-12-04 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Urinary Bladder, Overactive
Keywords: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Solifenacin Succinate; Tolterodine Tartrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Experimental): Solifenacin succinate 5/10mg
  Interventions: Drug: Solifenacin succinate
- II (Experimental): Tolterodine 4mg
  Interventions: Drug: Tolterodine

INTERVENTIONS:
Drug: Solifenacin succinate — oral
  Other Names: YM905; Vesicare
  Arms: I
Drug: Tolterodine — Oral
  Arms: II

SUMMARY:
Prospective, double-blind, double-dummy, 2-arm, parallel-group, design. Flexible dose regimen for solifenacin succinate, fixed dose treatment regimen for tolterodine. Assessment of OAB symptoms by patient diaries.

ELIGIBILITY:
Inclusion Criteria:

At study entry:

* Patient is willing and able to complete the micturition diary correctly
* Symptoms of overactive bladder (including urinary frequency, urgency or urge incontinence) for >= 3 months

At randomization:

* Patient must experience frequency of micturition on average >= 8 times per 24 hour period during the 3 day micturition diary period
* Patient must experience at least one of the following symptoms during the 3 day micturition diary period:

  * At least 3 episodes of urinary incontinence or,
  * Patients must exhibit urgency at least 3 times

Exclusion Criteria:

At study entry:

* Pregnant women or women who intend to become pregnant during the study or women of childbearing potential who are sexually active and practising an unreliable method of birth control or will be lactating during the study. Reliable contraceptive methods are intra-uterine devices, contraceptive pills of combination type, hormonal implants and injectable contraceptives
* Clinically significant outflow obstruction (at the discretion of the investigator)
* Significant post void residual volume (PVR>200ml)
* Significant stress incontinence or mixed stress/urge incontinence where stress is the predominant factor as determined by the investigator
* Patient with a neurological cause for abnormal detrusor activity
* Evidence of a symptomatic urinary tract infection, chronic inflammation such as interstitial cystitis, bladder stones, previous pelvic radiation therapy or previous or current malignant disease of the pelvic organs
* Uncontrolled narrow angle glaucoma, urinary or gastric retention or any other medical condition which in the opinion of the investigator makes the use of anticholinergics contra-indicated
* Non drug treatment including electrostimulation therapy or start of a bladder training program during the 2 weeks prior to entry into, or during the study
* Use of drugs intended to treat urinary incontinence
* Diabetic neuropathy
* Known or suspected hypersensitivity to solifenacin, tolterodine, other anticholinergics or lactose
* Any clinically significant condition, which in the opinion of the investigator makes the patient unsuitable for the trial
* Participation in any clinical trial within 30 (90 in the UK) days prior to randomisation
* Employees of the Yamanouchi Group, third parties associated with the study, or the study site

At randomization:

* Patient who did not complete the micturition diary according to the instructions
* Total daily urine volume > 3000 ml as verified in the micturition diary

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1355 (Actual)
Dates: Start 2003-07; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean number of micturitions per 24 hours | Weeks 4, 8 and 12

SECONDARY OUTCOMES:
Change from baseline in mean urgency frequency per 24 hours | Weeks 4, 8 and 12
Change from baseline in mean number of incontinence and urge incontinence episodes per 24 hours | Weeks 4, 8 and 12
Change from baseline in mean volume voided per micturition | Weeks 4, 8 and 12
Change from baseline in number of pads used | Weeks 4, 8 and 12
Change from baseline in mean nocturia episodes per 24 hours | Weeks 4, 8 and 12
Percentage of patients requiring an increase in the dose of the study medication | Weeks 4, 8 and 12
Change from baseline in patient perception of bladder condition | Weeks 4, 8 and 12
Patient assessment of treatment benefit | Weeks 4, 8 and 12
Physician assessment of treatment benefit | Weeks 4, 8 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Chair — Astellas Pharma Europe B.V.
Locations (95):
- Minsk, Belarus
- Belgium (4):
  - Antwerp
  - Brussels
  - Ghent
  - Middleheim
- Czechia (5):
  - Brno
  - Bulovce
  - České Budějovice
  - Mělník
  - Prague
- Denmark (7):
  - Aalborg
  - Aarhus
  - Copenhagen
  - Glostrup Municipality
  - Herlev
  - Kolding
  - Odense
- France (10):
  - Angers
  - Bordeaux
  - Clermont-Ferrand
  - Lille
  - Nantes
  - Paris
  - Reims
  - Rouen
  - Saint-Priest-en-Jarez
  - Toulouse
- Germany (10):
  - Bad Ems
  - Emmendingen
  - Frankfurt
  - Freiburg im Breisgau
  - Hagenow
  - Hamburg
  - Koblenz
  - Rheinfelden
  - Trier
  - Uetersen
- Greece (4):
  - Athens
  - Larissa
  - Pátrai
  - Thessaloniki
- Hungary (4):
  - Budapest
  - Nyíregyháza
  - Szolnok
  - Tatabánya
- Italy (8):
  - Montecchio Emilia
  - Novara
  - Orbassano
  - Rome
  - Sassari
  - Sesto San Giovanni
  - Varese
  - Verona
- Netherlands (8):
  - Apeldoorn
  - Ede
  - Eindhoven
  - Groningen
  - Nijmegen
  - Roermond
  - Tilburg
  - Zeist
- Norway (4):
  - Bodø
  - Haugesund
  - Rud
  - Tønsberg
- Russia (2):
  - Moscow
  - Saint Petersburg
- Slovakia (5):
  - Bratislava
  - Košice
  - Martin
  - Prešov
  - Skalica
- Spain (9):
  - Alicante
  - Bilbao
  - Burgos
  - Llobregat
  - Madrid
  - Santiago de Compostela
  - Seville
  - Valencia
  - Valladolid
- Sweden (4):
  - Gothenburg
  - Malmo
  - Nyköping
  - Stockholm
- Kiev, Ukraine
- United Kingdom (9):
  - Birmingham
  - Harrow
  - Leicester
  - Liverpool
  - London
  - Plymouth
  - Sheffield
  - Stevenage
  - Swansea

REFERENCES:
- [Background] Chapple CR, Martinez-Garcia R, Selvaggi L, Toozs-Hobson P, Warnack W, Drogendijk T, Wright DM, Bolodeoku J; STAR study group. A comparison of the efficacy and tolerability of solifenacin succinate and extended release tolterodine at treating overactive bladder syndrome: results of the STAR trial. Eur Urol. 2005 Sep;48(3):464-70. doi: 10.1016/j.eururo.2005.05.015. PMID 15990220